CLINICAL TRIAL: NCT04094545
Title: Intestinal Flora Disruption and a Novel Intestinal Biomarker Associated With Nasopharyngeal Carcinoma
Brief Title: Intestinal Flora Sequencing for Nasopharyngeal Carcinoma
Status: Completed | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: ThirdXiangyaJHY
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2018-09

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Biomarker; nasopharyngeal carcinoma; familial; sporadic; intestinal flora
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The faeces and the sera of the recruited participants
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nasopharyngeal carcinoma(NPC): The patients (1) were diagnosed with NPC; 2)18< Age <75.
- Health adults: (1) 18< Age <75, and Han Chinese residents living in Hunan more than 3 years. (2) Health examination population who physical examination, assistant examination and serological examination were normal; None of the patients had rhinitis or used any antibiotics during the three months last 3 months.

SUMMARY:
This study investigated the correlation between the changes in the intestinal flora and NPC by an examination of the intestinal flora and multiple clinical indicators of the blood of 8 carefully screened patients of familial NPC, 24 patients of sporadic NPC and 27 healthy controls and a comparison of the differences in their intestinal flora structures and biological functions. By analyzing the function of the intestinal floras of NPC patients, we aimed to provide a better biological marker for patients with familial and sporadic NPC and constructed a disease prediction model for high-risk populations.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is a malignant nasopharyngeal disease with a complicated etiology that occurs mostly in southern China. Intestinal flora imbalance is believed to be associated with a variety of organ malignancies. Currently, the relationship between intestinal flora and NPC is not clear, although many studies have shown that intestinal flora can be used as a biomarker for many cancers and to predict cancer.

To compare the differences in intestinal flora compositions and biological functions among patients with familial NPC (NPC_F), patients with sporadic NPC (NPC_S) and healthy controls (NOR), we compared the intestinal flora DNA sequencing and hematological testing results between every two groups using bioinformatic methods.

ELIGIBILITY:
Inclusion Criteria:

* NPC patients with a first degree family history of NPC
* NPC patients without any kind of tumor family history

Exclusion Criteria:

* Informed refusal.
* Lack of necessary tests and patient test information is not detailed

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We recruited 481 NPC patients and staged their tumor status with the AJCC 7th edition staging criteria，at the same time, 87 healthy volunteers were recruited.
Sampling Method: Probability Sample
Enrollment: 568 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
family NPC patients | through study completion, an average of 1 year
  NPC patients with a first degree NPC family history
sporadic NPC patients | through study completion, an average of 1 year
  NPC patients without any tumor family history

CONTACTS AND LOCATIONS:
Locations (1):
- the Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bei JX, Li Y, Jia WH, Feng BJ, Zhou G, Chen LZ, Feng QS, Low HQ, Zhang H, He F, Tai ES, Kang T, Liu ET, Liu J, Zeng YX. A genome-wide association study of nasopharyngeal carcinoma identifies three new susceptibility loci. Nat Genet. 2010 Jul;42(7):599-603. doi: 10.1038/ng.601. Epub 2010 May 30. PMID 20512145
- [Result] Bhatt AP, Redinbo MR, Bultman SJ. The role of the microbiome in cancer development and therapy. CA Cancer J Clin. 2017 Jul 8;67(4):326-344. doi: 10.3322/caac.21398. Epub 2017 May 8. PMID 28481406
- [Result] Bokulich NA, Kaehler BD, Rideout JR, Dillon M, Bolyen E, Knight R, Huttley GA, Gregory Caporaso J. Optimizing taxonomic classification of marker-gene amplicon sequences with QIIME 2's q2-feature-classifier plugin. Microbiome. 2018 May 17;6(1):90. doi: 10.1186/s40168-018-0470-z. PMID 29773078
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Chung H, Pamp SJ, Hill JA, Surana NK, Edelman SM, Troy EB, Reading NC, Villablanca EJ, Wang S, Mora JR, Umesaki Y, Mathis D, Benoist C, Relman DA, Kasper DL. Gut immune maturation depends on colonization with a host-specific microbiota. Cell. 2012 Jun 22;149(7):1578-93. doi: 10.1016/j.cell.2012.04.037. PMID 22726443
- [Result] Escobar JS, Klotz B, Valdes BE, Agudelo GM. The gut microbiota of Colombians differs from that of Americans, Europeans and Asians. BMC Microbiol. 2014 Dec 14;14:311. doi: 10.1186/s12866-014-0311-6. PMID 25495462
- [Result] Ferlay J, Colombet M, Soerjomataram I, Mathers C, Parkin DM, Pineros M, Znaor A, Bray F. Estimating the global cancer incidence and mortality in 2018: GLOBOCAN sources and methods. Int J Cancer. 2019 Apr 15;144(8):1941-1953. doi: 10.1002/ijc.31937. Epub 2018 Dec 6. PMID 30350310
- [Result] Goodrich JK, Waters JL, Poole AC, Sutter JL, Koren O, Blekhman R, Beaumont M, Van Treuren W, Knight R, Bell JT, Spector TD, Clark AG, Ley RE. Human genetics shape the gut microbiome. Cell. 2014 Nov 6;159(4):789-99. doi: 10.1016/j.cell.2014.09.053. PMID 25417156